CLINICAL TRIAL: NCT02909101
Title: Cognitive Training to Reduce Impulsivity in HIV-infected Cocaine Users
Brief Title: Project IMPACT: Improving Memory Performance by Applying Cognitive Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00053630_1
Record Dates: First submitted 2016-09-16; First posted 2016-09-21 (Estimated); Results first posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Cocaine Use Disorders; HIV
Keywords: Working memory; cognitive training; HIV; substance abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active Cognitive Training (ACT) (Experimental): Participants will complete computerized games designed to enhance working memory. Participants will complete 48 training sessions over 8 weeks.
  Interventions: Device: Active Cognitive Training (ACT)
- Control Training (CON) (Sham Comparator): Participants will complete 48 training sessions over 8 weeks. The control games are not designed to enhance memory.
  Interventions: Device: Control Training (CON)

INTERVENTIONS:
Device: Active Cognitive Training (ACT) — Cognitive training games
  Other Names: Lumosity
  Arms: Active Cognitive Training (ACT)
Device: Control Training (CON) — Cognitive training games
  Other Names: Lumosity
  Arms: Control Training (CON)

SUMMARY:
The purpose of this study is to examine the effects of a cognitive training program in persons with Human Immunodeficiency Virus (HIV) infection who have used cocaine. This study tests the feasibility and preliminary efficacy of a computerized cognitive training program to improve working memory and decrease impulsivity (delay discounting) among HIV-infected individuals.

DETAILED DESCRIPTION:
Of the 1.2 million Americans living with HIV, over half experience neurocognitive impairments (NCI) that adversely affect daily living and are predictive of increased morbidity and mortality. HIV-infected individuals who are addicted to stimulant drugs like cocaine are at even higher risk for NCI, which contributes to impulsive decision making, and engage in high rates of risky behaviors that are associated with both poor clinical outcomes and HIV transmission to others. Delay discounting, a key aspect of impulsivity, describes the tendency to devalue a reward as the delay to its receipt increases. Individuals addicted to drugs tend to prefer smaller, immediate rewards over larger, delayed rewards. Excessive discounting is associated with a wide range of other health risk behaviors, including risky sex. The Competing Neurobehavioral Decision Systems model posits that excessive discounting results from greater relative strength of the impulsive system over the executive control system. The investigators' own work suggests that HIV infection modulates the effect of cocaine on brain functioning in the executive control network during delay discounting. Prior research supports a robust association between excessive discounting and working memory impairment. As a core executive function that supports self-regulation, working memory is theoretically an intervention target for HIV risk reduction. Computerized working memory training has been shown to decrease delay discounting in stimulant users, but it has not yet been tested in HIV-infected drug users. The proposed R21 study will test the preliminary efficacy of a computerized cognitive training program to improve working memory and reduce delay discounting in HIV-infected cocaine users. Using a randomized trial design, the investigators will assign 50 participants to either the experimental cognitive training condition or an attention-matched control condition. Participants will complete 48 sessions in 8 weeks, with assessments at baseline, post-training, and 1-month follow-up to evaluate intervention effects. The investigators hypothesize that cognitive training will, relative to the control condition, lead to greater improvements in working memory and reductions in delay discounting. The investigators will also examine change in HIV risk behaviors (cocaine use, risky sex, and medication adherence). Results will support an R01 application for a larger scale trial to rigorously test the impact of cognitive training on HIV-related behavioral and clinical outcomes. This innovative line of research has important translational implications for HIV clinical practice, including dissemination in resource-limited settings with few neuropsychology specialists. This proposal directly advances a high priority topic for AIDS-designated funding by testing a novel treatment for HIV-associated NCI in drug users. By focusing on a high-risk population that continues to drive HIV transmission, this research has strong potential to improve neurobehavioral functioning in HIV-infected persons, and ultimately to reduce the incidence of new HIV infections.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* currently on antiretroviral medications for >3 months
* cocaine use as defined by crack/cocaine use in the past month, cocaine-type stimulant use disorder, and cocaine as the principal substance of abuse
* working memory impairment as defined by scoring >1 standard deviation below the normative mean on at least 2 out of the 3 working memory tests

Exclusion Criteria:

* pregnancy
* English non-fluency or illiteracy
* <8th grade education
* serious neurological disorders including HIV dementia, traumatic brain injury, severe mental illness, or acute psychiatric distress
* impaired mental status
* individuals who state they are planning to move away from the area within the next 3 months
* individuals without stable housing

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-02-23 (Actual); Study Completion 2019-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina S. Meade, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Cognitive Training (ACT): Participants will complete computerized games designed to enhance working memory. Participants will complete 48 training sessions over 10 weeks.
  Active Cognitive Training (ACT): Cognitive training games
- Control Training (CON): Participants will complete 48 training sessions over 10 weeks. The control games are not designed to enhance memory.
  Control Training (CON): Cognitive training games
Period: Overall Study
Arm/Group | Active Cognitive Training (ACT) | Control Training (CON)
Started | 29 | 29
Completed | 28 | 28
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Cognitive Training (ACT) | Control Training (CON) | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 29 | 58
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.97 (10.09) | 48.28 (8.28) | 48.62 (9.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 12 | 17
  Male | 24 | 17 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 29 | 29 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 24 | 50
  White | 1 | 3 | 4
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 29 | 58
Wechsler Test of Adult Reading (WTAR) [Mean (Standard Deviation); unit: units on a scale] — A word reading test that estimates premorbid verbal Intelligence Quotient (IQ). An intelligence quotient is a total score derived from several standardized tests designed to assess human intelligence. The WTAR comprises 50 words with irregular pronunciations that participants read aloud. The raw score on the WTAR ranges from 0 to 50. The raw score is transformed to an age-adjusted standard score (range 50-134), which is on the same scale as a full IQ test (M = 100; SD = 15). The age-adjusted standard WTAR score is used to provide an estimate for the full-scale IQ and is reported here.
  units on a scale | 81.97 (14.47) | 83.14 (13.75) | 82.55 (14.00)

OUTCOME MEASURES:

1. Primary Outcome: Working Memory Assessed by Domain Deficit Score
Description: Measured by domain deficit score, which is a continuous measure of overall impairment on the domain. 0 means no impairment and 5 means highest possible impairment.
Time Frame: Baseline; post-training, approximately 8 weeks
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Active Cognitive Training (ACT) | Control Training (CON)
Number analyzed (Participants) | 28 | 28
Score on a scale
  Baseline | .29 (.09) | .21 (.09)
  Post-training | .14 (.07) | .26 (.07)
Statistical Analysis 1: Comparison: Active Cognitive Training (ACT) vs Control Training (CON); Estimated marginal means, adjusted for covariates in the model, are reported. The p-value reported is for the Arm by Time interaction effect; Test type: Superiority; p = 0.039, ANCOVA; ANCOVAs were 2 (Arm) by 2 (Time). Covariates were age, WTAR standard score, and number of games improved (as a proxy of intervention engagement)

2. Secondary Outcome: Delay Discounting, Measured by the Monetary Choice Questionnaire (MCQ)
Description: The Monetary Choice Questionnaire (MCQ) is a standardized delay discounting task. Because scores are on a logarithmic scale, they were rank ordered for analysis. Ranks range from 1 to 13, with higher ranks meaning higher impulsivity.
Time Frame: Baseline; post-training, approximately 8 weeks
Population: One participant from ACT and two participants from CON were excluded because they did not provide valid responses on the MCQ at the post-training follow-up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Cognitive Training (ACT) | Control Training (CON)
Number analyzed (Participants) | 27 | 26
score on a scale
  Baseline | 8.70 (.41) | 7.97 (.42)
  Post-training | 8.38 (.37) | 8.76 (.38)
Statistical Analysis 1: Comparison: Active Cognitive Training (ACT) vs Control Training (CON); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.054, ANCOVA; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Acceptability as Measured by Participant Ratings
Description: Participants rated how satisfied they found the intervention on a 5 point scale (with 1 being very dissatisfied and 5 being very satisfied). Acceptability was defined a priori of achieving a mean rating of >3.5 on the 5 point scale.
Time Frame: Post-training, approximately 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Cognitive Training (ACT) | Control Training (CON)
Number analyzed (Participants) | 28 | 28
score on a scale | 4.04 (1.32) | 4.14 (1.11)
Statistical Analysis 1: Comparison: Active Cognitive Training (ACT) vs Control Training (CON); To determine acceptability, we examined whether mean ratings for both arms were above 3.5, and we also examined whether there was any difference between arms; Test type: Other; p = 0.744, t-test, 2 sided

4. Secondary Outcome: Acceptability as Measured by Participant Perception of Benefits and Barriers to Completing Sessions
Description: Participants rated how helpful they found the intervention on a 5 point scale (with 1 being very unhelpful and 5 being very helpful). Acceptability was defined a priori of achieving a mean rating of >3.5 on the 5 point scale for helpfulness.
Time Frame: Post-training, approximately 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Cognitive Training (ACT) | Control Training (CON)
Number analyzed (Participants) | 28 | 28
score on a scale | 4.14 (1.15) | 4.04 (1.02)
Statistical Analysis 1: Comparison: Active Cognitive Training (ACT) vs Control Training (CON); To determine acceptability in terms of helpfulness, we examined whether mean ratings for both arms were above 3.5, and we also examined whether there was any difference between arms; Test type: Other; p = 0.719, t-test, 2 sided

5. Secondary Outcome: Percent Medication Adherence Across All Antiretroviral Medications
Description: 0% indicates no doses of medications were taken, and 100% means all doses were taken.
Time Frame: Baseline; post-training, approximately 8 weeks
Measure: Mean (Standard Error); unit: percentage of doses
Arm/Group | Active Cognitive Training (ACT) | Control Training (CON)
Number analyzed (Participants) | 28 | 28
percentage of doses
  Baseline | 96.53 (2.29) | 88.97 (2.29)
  Post-training | 96.08 (2.19) | 92.03 (2.19)
Statistical Analysis 1: Comparison: Active Cognitive Training (ACT) vs Control Training (CON); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.337, ANCOVA; [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Sexual Risk Behavior as Measured by the Risk Assessment Battery (RAB)
Description: The RAB is a standardized survey. Scores range from 0 to 18, with higher scores meaning greater sexual risk.
Time Frame: Baseline; post-training, approximately 8 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Cognitive Training (ACT) | Control Training (CON)
Number analyzed (Participants) | 28 | 28
score on a scale
  Baseline | 4.53 (.43) | 3.68 (.43)
  Post-training | 4.04 (.47) | 4.21 (.47)
Statistical Analysis 1: Comparison: Active Cognitive Training (ACT) vs Control Training (CON); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.025, ANCOVA; [statistical method as in outcome 1, analysis 1]

7. Secondary Outcome: Number of Days of Cocaine Use as Measured by Timeline Followback Interview Methodology
Description: The Timeline Followback Method involves asking subjects to retrospectively estimate their cocaine use 30 days prior to the interview date. Responses therefore range from 0 to 30 days.
Time Frame: Baseline; post-training, approximately 8 weeks
Measure: Mean (Standard Error); unit: days
Arm/Group | Active Cognitive Training (ACT) | Control Training (CON)
Number analyzed (Participants) | 28 | 28
days
  Baseline | 7.51 (1.68) | 6.88 (1.68)
  Post-training | 8.49 (1.72) | 5.12 (1.72)
Statistical Analysis 1: Comparison: Active Cognitive Training (ACT) vs Control Training (CON); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.133, ANCOVA; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Approximately 17 weeks (from Baseline to the follow-up assessment)
Arm/Group | Active Cognitive Training (ACT) | Control Training (CON)
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT02909101/Prot_SAP_000.pdf